CLINICAL TRIAL: NCT05525858
Title: KOrean Precision Medicine Networking Group Study of MOlecular Profiling Guided Therapy Based on Genomic Alterations in Advanced Solid Tumors II
Brief Title: KPMNG Study of MOlecular Profiling Guided Therapy Based on Genomic Alterations in Advanced Solid Tumors II
Acronym: KOSMOSII
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Korean Cancer Study Group (Other); Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Jee Hyun Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: KCSG AL 22-09
Record Dates: First submitted 2022-08-29; First posted 2022-09-02 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor; Advanced Solid Tumor; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — alectinib; atezolizumab; Erlotinib Hydrochloride; Trastuzumab; pertuzumab; Ado-Trastuzumab Emtansine; Vemurafenib; Bevacizumab; entrectinib; pralsetinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Patients who have insufficient genomic information from their NGS results (e.g., lack of variant calling format file or uninterpretable reports) or who are candidates of immunotherapy will submit their tissue and/or blood, for central NGS testing and exploratory biomarker analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tier 1. Therapeutic use of investigational products (KOSMOS-II drugs): If there are no drugs available under current regulation or patients are not feasible to any clinical trials, and If tumors have actionable genetic alterations and approved drug in any indications but tumor type is not indicative, the MTB may recommend one of KOSMOS-II drugs, therapeutic use of investigational products.
  Interventions: Drug: Alectinib; Drug: Atezolizumab; Drug: Erlotinib; Drug: Trastuzumab + Pertuzumab; Drug: Trastuzumab emtansine; Drug: Vemurafenib; Drug: Bevacizumab + Erlotinib; Drug: Entrectinib; Drug: Pralsetinib
- Tier 2: Alternative treatments: If there are no KOSMOS-II drugs (Tier 1) or clinical trials (Tier 3) appropriate for patients, the MTB may recommend alternative treatment options (e.g., conventional therapy, radiotherapy, or supportive care).
- Tier 3: Clinical trial: If patient is eligible for clinical trials matched for actionable genomic alterations found in NGS testing, the MTB will recommend enrollment to clinical trials.

INTERVENTIONS:
Drug: Alectinib — ALK fusion or mutations, Mutations or amplification in any of the following: RET
  Other Names: Alecensa
  Groups: Tier 1. Therapeutic use of investigational products (KOSMOS-II drugs)
Drug: Atezolizumab — MSI high status by any method Or Any mutation in any of these genes:
  MLH1 or MSH2 or MSH6 or PMS2 or EPCAM Or Any of the following mutations in POLE: R150X, P286R, P286H, S297F, Y298fs, F367S, V411, L424V, P436R, S459F, R665W, L698fs, R762W, R1519C, R1826W, D316H, D316G, R409W, L474P Or Any of the following mutations in POLD1: P112fs, A930fs, S478N Or Any mutation in the following: POLE not listed above, POLD1 not listed above, POLD2, POLD3, POLD4, POLQ or PRKDC Or Any loss of function mutations in BRCA1, BRCA2, ATM, MSH3, PMS1, MLH3, EXO1, RFC1, RFC2, RFC3, RFC4, RFC5, PCNA, RPA1, PRA2, PRA3, PRA4, or SSBP1 High tumor mutational burden decided by KOSMOS-II MTB (TMB ≥20/Mb in local NGS or if 10-20/Mb, confirmed by central NGS te sting)
  Other Names: Tecentriq
  Groups: Tier 1. Therapeutic use of investigational products (KOSMOS-II drugs)
Drug: Erlotinib — EGFR Exon 19 deletions in the region E746_E759;
  Any of the following EGFR mutations:
  E709A, E709G, E709K, E884K, G719A, G719C, G719S, L858R, L861Q, L833V, S768I
  Other Names: Tarceva
  Groups: Tier 1. Therapeutic use of investigational products (KOSMOS-II drugs)
Drug: Trastuzumab + Pertuzumab — ERBB2 amplification, or over-expression; or presence of any of the following ERBB2 mutations:
  G309A, G309E, S310F, S310Y, R678Q, I655V, D769H, D769Y, L755S, p.L75 5_T759del, I767M, V777L, E321G, R896C; P780ins; delL755-T759 ERBB2 amplification or approved by the KOSMOS Molecular Tumor Board
  Other Names: Herceptin + Perjeta
  Groups: Tier 1. Therapeutic use of investigational products (KOSMOS-II drugs)
Drug: Trastuzumab emtansine — ERBB2 amplification, or over-expression; or presence of any of the following ERBB2 mutations:
  G309A, G309E, S310F, S310Y, R678Q, I655V, D769H, D769Y,L755S, p.L75 5_T759del, I767M, V777L, E321G, R896C; P780ins; delL755-T759 ERBB2 oncogenic mutations; G152V, X215_splice, D277Y, G292C, N302K, V308M, G309A, S310F, S310Y, S244C, L651V, V659E, G660D, R678Q, V697L, G727A, T733I, L755A, L755P, L755S, D769H, D769Y, A775_G776insSVMA, A775_G776insYVMA (i.e.,Y772_A775dup,M774_A775insAYVME 770delinsEAYVM), G776_V777 > AVCV, G776_V777 > AVGCV, G776_V777 > VCV, G776_V777insVC, G776C, G776delinsLCT, G776L, G776dleinsVC, G776L777_G778insC, V777L, V777M, G778_Y779insGSP, P780_Y781insGSP (i.e.,G778_P780dup), L786V, N813D, R840W, V842I, T862A, R896G, E1021Q or approved by the KOSMOS Molecular Tumor Board
  Other Names: Kadcyla
  Groups: Tier 1. Therapeutic use of investigational products (KOSMOS-II drugs)
Drug: Vemurafenib — BRAF_V600E/D/K/R mutations
  Other Names: Zelboraf
  Groups: Tier 1. Therapeutic use of investigational products (KOSMOS-II drugs)
Drug: Bevacizumab + Erlotinib — FH inactivating mutations or approved by the KOSMOS Molecular Tumor Board
  Other Names: Avastin + Tarceva
  Groups: Tier 1. Therapeutic use of investigational products (KOSMOS-II drugs)
Drug: Entrectinib — ROS1 gene fusion using either a fluo rescence in situ hybridization (FISH) or next-generation sequencing (NGS) or approved by the KOSMOS Molecular Tumor Board
  Other Names: Rozlytrek
  Groups: Tier 1. Therapeutic use of investigational products (KOSMOS-II drugs)
Drug: Pralsetinib — RET fusion or mutations; CCDC6 RET, RET V804L, RET V804M, RET M918T, KIF5B-RET, RET C634W or approved by the KOSMOS Molecular Tumor Board
  Other Names: Gavreto
  Groups: Tier 1. Therapeutic use of investigational products (KOSMOS-II drugs)

SUMMARY:
A national, prospective, multi-center, open-label, multi-cohort study comprised of a framework to screen patients for actionable targets and evaluation of molecular profiling guided therapy recommended by MTB based on genomic alterations using targeted and/or immunotherapies outside of the approved indications via local clinical practice (Tier 1 & 2) and clinical trials (Tier 3)

DETAILED DESCRIPTION:
A. The KOSMOS-II study will recruit locally advanced or metastatic solid tumor patients who had disease progression on standard first line anti-cancer treatment and/or has no standard treatment option, in order to prove MTB value to guide treatment within local clinical practice.

B. After site physicians confirm that NGS results of patients are available, they preliminarily decide initial treatment before MTB submission and collect informed consent form, and then patients can register to the KOSMOS-II study. Site physicians upload patients' clinical, pathologic, and genomic data for MTB submission. If site physician cannot determine initial treatment before MTB, site physician can record 'initial treatment cannot be determined' and can register the patient for MTB.

C. MTB records its treatment recommendations within available drugs list based on uploaded data, then site physicians make a final treatment decision, after informing patient about MTB decision and assessment of patients' final health status and preference.

D. Patients who have insufficient genomic information from their NGS results (e.g., lack of variant calling format file or uninterpretable reports) or who are candidates of immunotherapy will submit their tissue and/or blood, for central NGS testing and exploratory biomarker analysis.

E. Recommended treatment option There are three different options including (1) Tier 1: Therapeutic use of investigational products (KOSMOS-II drugs), (2) Tier 2: alternative treatment options, and (3) Tier 3: clinical trials

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Histologically proven locally advanced or metastatic solid tumors*** who showed disease progression on standard first line anti-cancer treatment and/or has no standard treatment option

  *** very rare diseases without standard treatment option which form solid mass, such as Erdheim Chester disease can be enrolled after KOSMOS MTB approval
* A genomic test results must be available in a MFDS-accredited for laboratories offering service, or in part of clinical trial/study or other commercial labs approved and certified by regulatory bodies compatible with MFDS, such as CLIA. A genomic test can be conducted with tumor tissue as well as plasma circulating tumor DNA.

  1. Results from genomic profiling tests performed after diagnosis with metastatic/advanced disease to registration are acceptable. NGS results performed within three years prior to registration are preferred. Those patients with NGS results from primary tumor or more than 3 years prior to enrollment can be registered and whether NGS data is acceptable will be subject to MTB decision.
  2. NGS panels should be i. Tested in a lab that is accredited by one or more quality assurance program (e.g., Korean Institute of Genomic Testing Evaluation, The Korean Society of Pathologists, Korean Society for Laboratory Medicine, Korea Laboratory Accreditation Scheme, etc.) ii. Patients who have insufficient genomic information from their NGS results (e.g., lack of variant calling format file or uninterpretable reports) or who are candidates of immunotherapy will submit their tissue and/or blood, for central NGS testing and exploratory biomarker analysis.
* Ability to understand and the willingness to sign a written informed consent document
* Life expectancy of at least 12 weeks
* Adequate recovery from most recent systemic or local treatment for cancer.

Exclusion Criteria:

* Patients receiving any anti-cancer treatment (local treatment, chemotherapy, immunotherapy, targeted therapy) within 2 weeks prior to the start of study treatment
* Any clinical condition, according to the opinion of site physicians, which makes molecular profiling guided therapy not at the best interest of the participating patient.
* Patients who have ongoing toxicities of ≥ CTCAE 2, other than peripheral neuropathy, related to previous anti-cancer treatment. Patients with ongoing peripheral neuropathy of ≥ CTCAE 3 will be excluded. Laboratory abnormalities ≥ CTCAE 2 considered as not clinically significant by the study physician will be allowed.
* Pregnant or breastfeeding, or intending to become pregnant during the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically proven locally advanced or metastatic solid tumor patients with disease progression on standard first line anti-cancer treatment and/or has no standard treatment option
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of molecular profiling guided therapies (MGT) based on genomic alterations in patients with advanced solid tumors in terms of the proportion of receipt of the treatment | 12 months after treatment initiation (estimated average)
  Percentage of patients who receive molecular profiling guided therapy as recommended by MTB, either in therapeutic use of investigational products (KOSMOS-II drugs), alternative treatment, or clinical trial.
To evaluate the effectiveness of molecular profiling guided therapies in terms of clinical benefit rate (CR/PR/SD beyond 16 +/- 2 weeks) in Tier 1* population | Assessed at 16 weeks of treatment
  Percentage of patients achieving response defined as CR/PR/SD at 16 ± 2 weeks reported by site physician

SECONDARY OUTCOMES:
Objective response rate | 12 months after treatment initiation (estimated average)
  The proportion of patients who obtained CR/PR as the best response according to the RECIST 1.1 criteria
Progression-free survival | 12 months after treatment initiation (estimated average)
  Progression-free survival in accordance with local clinical practice
Treatment duration | 12 months after treatment initiation (estimated average)
  The period from the start of treatment to the end of treatment for any reason
1-year overall survival rate | 12 months after treatment initiation (estimated average)
  Proportion of patients alive 1 year after study registration
To evaluate safety of molecular profiling guided therapies | 12 months after treatment initiation (estimated average)
  The incidence of serious adverse events will be calculated among the adverse events in patients with Tier 1 and Tier 3. ( based on NCI-CTCAE v5.0 )

CONTACTS AND LOCATIONS:
Overall Officials: JEEHYUN KIM, Study Director — Seoul National University Bundang Hospital
Locations (32):
- South Korea (32):
  - Soonchunhyang University Hospital Bucheon, Bucheon-si
  - Chungbuk National University Hospital, Chungju
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang
  - Chonnam National University Hwasun Hospital, Hwasun
  - Gachon University Gil Medical Center, Incheon
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Dong-A University Hospital, Pusan
  - Cha University Bundang Medical Center, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Chung-ang University Hospital, Seoul
  - Ewha womans university Mokdong Hospital, Seoul
  - Gangbuk Samsung Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Yonsei Cancer Hospital, Seoul
  - Ajou University Hospital, Suwon
  - The Catholic University of Korea, ST. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan

REFERENCES:
- [Derived] Kim SY, Kim JH, Kim TY, Park SR, Yoon S, Lee S, Lee SH, Kim TM, Han SW, Kim HR, Yun H, Lee S, Kim J, Choi YL, Choi KS, Chae H, Ryu H, Lee GW, Zang DY, Ahn JB. Pragmatic nationwide master observational trial based on genomic alterations in advanced solid tumors: KOrean Precision Medicine Networking Group Study of MOlecular profiling guided therapy based on genomic alterations in advanced Solid tumors (KOSMOS)-II study protocol KCSG AL-22-09. BMC Cancer. 2024 May 9;24(1):574. doi: 10.1186/s12885-024-12338-y. PMID 38724991